CLINICAL TRIAL: NCT02909842
Title: Immunomodulating Effects of Drinking Fermented Milk Containing Lactobacillus Paracasei (IMULUSTM): a Randomized Controlled Trial Using an Influenza Vaccination Model
Brief Title: Effect of Drinking Fermented Milk on Immune Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Dunyaporn Trachootham, Assistant Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MU-CIRB 2015/145.2509
Record Dates: First submitted 2016-09-14; First posted 2016-09-21 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Influenza
Keywords: influenza; vaccine; probiotic; immune response
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Experimental): Seasonal Influenza Vaccine (H1N1, H3N2, PhuB) and 100 ml bottle of yoghurt drink, unlabelled drinking fermented milk containing probiotic, Lactobacillus paracasei (IMULUS)
  Interventions: Dietary Supplement: Drinking fermented milk; Biological: Seasonal Influenza Vaccine (H1N1, H3N2, PhuB)
- control group (Placebo Comparator): Seasonal Influenza Vaccine (H1N1, H3N2, PhuB) and 100 ml bottle of placebo, unlabelled acidified milk with similar physical and sensory appearance to the experimental one
  Interventions: Dietary Supplement: placebo; Biological: Seasonal Influenza Vaccine (H1N1, H3N2, PhuB)

INTERVENTIONS:
Dietary Supplement: Drinking fermented milk — Drinking fermented milk containing Lactobacillus paracasei (IMULUS)
  Arms: study group
Dietary Supplement: placebo — Acidified placebo milk with similar physical characteristics to the yoghurt drink
  Arms: control group
Biological: Seasonal Influenza Vaccine (H1N1, H3N2, PhuB) — Intramuscular injection of a single shot of influenza vaccine

SUMMARY:
This blinded randomized controlled trial aims to investigate the effect of drinking fermented milk containing Lactobacillus paracasei (IMULUS) on immune response against influenza.

DETAILED DESCRIPTION:
This study is conducted in healthy volunteer using product approved by Thai FDA. This blinded randomized controlled trial compare immune response against influenza H1N1, H3N2 and Phu-B between study group and control group. The study group receives influenza vaccine and drinking fermented milk containing Lactobacillus paracasei (IMULUS), while the control group receives influenza vaccine and placebo acidified milk. The trial lasts for 8 weeks and include four time points of data collection (0, 2, 6, 8 weeks). Subjects, outcome assessor and investigators are blinded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 45 years old
* healthy and having normal vital signs
* no history of uncontrolled systemic or autoimmune diseases
* no signs or symptoms of respiratory infection
* normal blood chemistry including complete blood count (CBC), liver and kidney function, lipid profile and fasting blood sugar
* no history of influenza vaccine during the past 6 months
* able to continuously take the intervention daily for 6 weeks
* able to refrain from other probiotic products such as drinking fermented milk or yoghurt since the beginning till the end of data collection
* accepted to receive influenza vaccine shot
* able to refrain from receiving other vaccine during the trial
* able to refrain from traveling to endemic area of influenza
* able to communicate in Thai and sign their written inform consent

Exclusion Criteria:

* under pregnancy or expected to be pregnant
* lactose or milk protein intolerances
* daily intake of probiotic product for one month prior to recruitment
* chronic alcoholism
* GI disturbance e.g. stomachache, frequent diarrhea or constipation
* history of GI surgery
* ongoing treatment with antibiotic or other immune affecting drugs e.g. glucocorticoids, chemotherapy, antibodies, ciclosporin, hormone and opioids

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-01; Primary Completion 2016-09-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Immune response rate for H1N1, H3N2 and Phu-B virus | 4 weeks after vaccination
  Number of subjects with increased HAI titer from baseline divided by total number of subjects

SECONDARY OUTCOMES:
Antibody response rate for influenza A (H1N1+H3N2) virus | 4 weeks after vaccination
  Number of subjects with increased Immunoglobulin G or M (IgG or IgM) antibody levels from baseline divided by total number of subjects
Changes from baseline immunoglobulin M (IgM) levels for influenza A (H1N1+H3N2) virus | 0, 2, 6 and 8 weeks after baseline
  Changes in serum levels of IgM antibody against influenza A, detected by ELISA assay
Changes from baseline immunoglobulin G (IgG) levels for influenza A (H1N1+H3N2) virus | 0, 2, 6 and 8 weeks after baseline
  Changes in serum levels of IgG antibody against influenza A, detected by ELISA assay
Changes from baseline HAI titer for H1N1, H3N2 and Phu-B virus | 0, 2, 6 and 8 weeks after baseline
  Changes in maximum dilution of serum, detected by Heme agglutination inhibition (HAI) assay , which can immunologically react against H1N1, H3N2 and Phu-B virus

CONTACTS AND LOCATIONS:
Overall Officials: Dunyaporn Trachootham, DDS, PhD, Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: No
Only summary of data will be reported. No individual data will be released.